CLINICAL TRIAL: NCT02333292
Title: Efficacy and Safety of Treatment Against Hepatitis C Virus Infection Based on Direct-acting Antivirals in Real-life Conditions: The GEHEP Cohort
Brief Title: Efficacy and Safety of Therapy Against HCV Based on Direct-acting Antivirals in Real-life Conditions
Acronym: FPSMON201401
Status: Completed | Type: Observational
Sponsor: Valme University Hospital (Other)
Collaborators: Hospital del SAS de Jerez (Other); Hospital General Universitario Elche (Other); Hospital La Línea de la Concepción (Unknown); Complexo Hospitalario Universitario de A Coruña (Other); Hospital de Figueres (Unknown); Hospital Universitario Puerto Real (Other); Hospital Universitario Virgen de la Victoria (Other); Hospital Universitario de Canarias (Other); Hospital General Universitario de Alicante (Other); Hospital Universitario Araba (Other); Hospital Royo Vilanova (Unknown); Hospital Universitario de Burgos (Other); Complejo Hospitalario Universitario de Huelva (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospital Universitario Virgen Macarena (Other); Complejo Hospitalario Universitario de Vigo (Other); Clinica Universidad de Navarra, Universidad de Navarra (Other); Hospital Clinico Universitario San Cecilio (Other); Hospital Universitario La Fe (Other); Hospital General Universitario de Valencia (Other); Hospital Universitario Infanta Leonor (Other); Hospital Universitario de Gran Canaria (Unknown); Hospital General Universitario Santa Lucía (Other); Centro Penitenciario Alicante 1 (Unknown); Hospital Regional Universitario Carlos Haya (Other); Hospital Virgen de la Luz (Other); Hospital General Universitario de Castellón (Other); Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, Karin Neukam, Dr, Valme University Hospital
Other Study IDs: GEHEP-MONO; GEHEP-001 (Other: SEIMC-GEHEP)
Record Dates: First submitted 2014-12-15; First posted 2015-01-07 (Estimated); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Chronic Hepatitis C Infection
MeSH Terms: interventions — telaprevir; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Sofosbuvir; Simeprevir; daclatasvir; ledipasvir; ombitasvir; dasabuvir; velpatasvir; elbasvir; grazoprevir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IFN: HCV-infected patients, pre-treated or treatment-naïve, who start a regimen containing pegylated interferon in combination with any DAA
  Interventions: Drug: Telaprevir; Drug: Boceprevir; Drug: Sofosbuvir; Drug: Simeprevir
- IFN-free: HCV-infected patients, pre-treated or treatment-naïve, who start a regimen containing one or more DAA
  Interventions: Drug: Sofosbuvir; Drug: Simeprevir; Drug: Daclatasvir; Drug: Ledipasvir; Drug: ritonavir-boosted Paritaprevir/ Ombitasvir; Drug: Dasabuvir; Drug: Velpatasvir; Drug: Elbasvir; Drug: Grazoprevir

INTERVENTIONS:
Drug: Telaprevir — Initiation of a regimen containing TVR
  Other Names: TVR
  Groups: IFN
Drug: Boceprevir — Initiation of a regimen containing BOC
  Other Names: BOC
  Groups: IFN
Drug: Sofosbuvir — Initiation of a regimen containing SOF
  Other Names: SOF
Drug: Simeprevir — Initiation of a regimen containing SMV
  Other Names: SMV
Drug: Daclatasvir — Initiation of a regimen containing DCV
  Other Names: DCV
  Groups: IFN-free
Drug: Ledipasvir — Initiation of a regimen containing LDV
  Other Names: LDV
  Groups: IFN-free
Drug: ritonavir-boosted Paritaprevir/ Ombitasvir — Initiation of a drug combination of PTV/OTV
  Other Names: PTV/OTV
  Groups: IFN-free
Drug: Dasabuvir — Initiation of a regimen containing DBV
  Other Names: DBV
  Groups: IFN-free
Drug: Velpatasvir — Initiation of a regimen containing VPV
  Other Names: VPV
  Groups: IFN-free
Drug: Elbasvir — Initiation of a regimen containing EBV
  Other Names: EBV
  Groups: IFN-free
Drug: Grazoprevir — Initiation of a regimen containing GZR
  Other Names: GZR
  Groups: IFN-free

SUMMARY:
Objectives: 1) To evaluate la proportion of hepatitic C virus (HCV)-monoinfected patients who show sustained virologic response (SVR) to treatment including direct-acting antivirals (DAAs) in the clinical practice in clinical units that treat infectious diseases and 2) to determine the frequency of adverse events, including those that are severe and/or cause treatment interruption, in DAA-based therapy in this setting.

Design: Multicentric, prospective post-authorised cohort study. Setting: Hospitals of the Hepatitis Study Group (GEHEP) of the Spanish Society of Infectious Diseases and Microbiology (SEIMC).

Study population: HCV-monoinfected patients that initiate DAA-based treatment outside clinical trials.

Variables: The primary efficacy outcome variable is the proportion of patients who reach undetectable HCV-RNA 12 weeks after the scheduled end of therapy (SVR12). The primary safety outcome variable is the percentage of subjects who discontinue therapy due to adverse events.

Statistical analysis: A descriptive study will be performed, as well as a double sensibility analysis of the frequency of SVR12 using both an intention-to-treat and an on-treatment approach. Those variables that are associated with SVR12 with a p-value <0.2 will be included in a logistic regression analysis in which SVR12 will be the dependent variable.

DETAILED DESCRIPTION:
The incidence of hepatic decompensations and mortality is reduced considerable in patients who achieve sustained virologic response (SVR) to therapy against hepatitis C virus (HCV) infection. With the arrival of direct-acting antivirals (AAD) against HCV, rates of SVR are significantly higher than what was achieved with pegylated interferon (peg-IFN) in combination with ribavirin (RBV). Therefore, AADs could have a high impact in this context. Therefore, triple therapy against HCV genotype 1 based on the first-generation protease inhibitors (PI) telaprevir (TVR) or boceprevir (BOC) plus peg-IFN/RBV became standard therapy in 2011 and SVR rates as high as 68%-75% were reached in treatment-naïve patients. In treatment-experienced subjects, retreatment with triple therapy resulted in higher SVR rates than what was observed with dual therapy alone, however, treatment success strongly depends on the previous response pattern. Unfortunately, combinations based on TVR or BOC are not well tolerated, treatments are complex, costs are high and pharmacological interactions are frequently observed.

The next generation of DAAs offers increased response rates and, furthermore, a better safety pattern than TVR or BOC. Additionally, the dosing of the newer DAAs is easier and more convenient, and pharmacological interactions of the newer DAAs are easier to manage or even not relevant. The FDA has approved the second-generation PI simeprevir, the HCV non-structural (NS) protein NS 5B inhibitor sofosbuvir, as well as the inhibitors of NS 5A daclatasvir and ledipasvir. Apart from a better efficacy, safety and convenience, these new DAAs are active against HCV genotypes other than 1. Finally, some of the new DAAs can be administered in interferon-free regimens and therefore offer treatment options for interferon-intolerant individuals or for those with a contraindication for peg-IFN. Therefore, in the near future, the vast majority of HCV monoinfected patients will be treated with a combination including a DAA. Currently, the main problem is the high cost of the DAAs challenging the health systems.

In spite of the positive prospect regarding response rates to DAAs, there are a number of questions to be answered as soon as possible. On the one hand, the information on efficacy and safety of the DAAs available to date is derived from clinical trials that do not reflect the circumstances of the clinical practice. In this context, clinical trials usually include a considerably low proportion of patients with certain characteristics, such as cirrhotics. Data from the French cohort CUPIC reveal that this subgroup shows a lower tolerability of TVR or BOC than that reported in pivotal clinical trials. In fact, data obtained from this cohort resulted in a change of treatment guidelines for HCV monoinfected patients published by the Spanish Agency of Medicines. On the contrary, there is evidence based on observations made within the expanded access program study HEP3002 that individuals with advanced fibrosis show a efficacy and safety profile when treated with triple therapy that is more similar to that observed in clinical trials than within the CUPIC cohort. Nevertheless, in this study, exclusion criteria and follow-up were comparable to what is applied in clinical trials. Therefore, the study population may not reflect exactly the patient profile seen in real-life.

Currently, information on the distinct aspects of treatment against HCV including DAAs under real-life conditions in Spain is scarce. Clinicians at the Infectious Diseases Units treat a high number of HCV monoinfected patients. These physicians are confronted with a patient population in which a history of drug abuse is predominant, the majority of the individuals having consumed injecting drugs, who frequently suffer psychiatric pathology and who receive concomitant therapy that cause problems regarding drug-drug interactions and adherence. Also, the HCV genotype distribution is different to what is observed in Hepatology Units, being the genotype 1a predominant as compared to 1b, 3 and 4. Taken into account what was mentioned above, these factors could cause different rates of SVR to DAAs, interruptions and voluntary drop-outs as compared to what has been reported, especially in the difficult-to-treat population.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* initiation of therapy including a direct-acting antiviral against HCV

Exclusion Criteria:

* HIV-infection
* unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV-infected patients who initiated treatment against HCV including a direct-acting antiviral
Sampling Method: Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients with Sustained Virological Response | 48 weeks
  Efficacy of treatment against hepatitis C virus infection based on direct-acting antivirals in real-life conditions as reflected in proportion of patients who achieve sustained virological response 12 weeks after end of therapy.
Number of Participants with Adverse Events | 48 weeks
  Safety of treatment against hepatitis C virus infection based on direct-acting antivirals in real-life conditions as reflected in the number of patients with adverse events.

SECONDARY OUTCOMES:
Identification of predictors of SVR | 48 weeks
Analyze efficacy and safety in patients that receive methadone maintenance therapy | 48 weeks
Analyze efficacy and safety according to previous treatment outcome | 48 weeks
Analyze efficacy and safety in patients with cirrhosis | 48 weeks
Evaluate impact of SVR on biological, elastographical and clinical parameters | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Karin I Neukam, Dr, Principal Investigator — Valme University Hospital
Locations (1):
- Valme University Hospital, Seville, Andalusia, Spain

REFERENCES:
- [Result] Mancebo M, Real LM, Mira JA, Recio E, Perez E, Monje-Agudo P, Merchante N, Macias J, Neukam K, Pineda JA. Changes in the response to treatment against chronic hepatitis C between 1999 and 2015: data from a prospective cohort. Eur J Gastroenterol Hepatol. 2016 Nov;28(11):1253-7. doi: 10.1097/MEG.0000000000000705. PMID 27415157
- [Result] Macias J, Monge P, Mancebo M, Merchante N, Neukam K, Real LM, Pineda JA. High frequency of potential interactions between direct-acting antivirals and concomitant therapy in HIV/hepatitis C virus-coinfected patients in clinical practice. HIV Med. 2017 Aug;18(7):445-451. doi: 10.1111/hiv.12471. Epub 2016 Nov 24. PMID 27882706
- [Result] Neukam K, Morano-Amado LE, Rivero-Juarez A, Macias J, Granados R, Romero-Palacios A, Marquez M, Merino D, Ortega E, Alados-Arboledas JC, Cucurull J, Omar M, Ryan-Murua P, Pineda JA; Grupo de Estudio de Hepatitis Virica, of the Sociedad Espanola de Enfermedades Infecciosas y Microbiologia Clinica: GEHEP-SEIMC and Grupo de Estudio de Hepatitis Virica, of the Sociedad Andaluza de Enfermedades Infecciosas y Microbiologia Clinica: HEPAVIR/Red de Investigacion en SIDA (RIS-HEP07). Liver stiffness predicts the response to direct-acting antiviral-based therapy against chronic hepatitis C in cirrhotic patients. Eur J Clin Microbiol Infect Dis. 2017 May;36(5):853-861. doi: 10.1007/s10096-016-2871-x. Epub 2016 Dec 21. PMID 28004322
- [Result] Pineda JA, Morano-Amado LE, Granados R, Macias J, Tellez F, Garcia-Deltoro M, Rios MJ, Collado A, Delgado-Fernandez M, Suarez-Santamaria M, Serrano M, Miralles-Alvarez C, Neukam K; Grupo de Estudio de Hepatitis Virica, of the Sociedad Espanola de Enfermedades Infecciosas y Microbiologia Clinica: GEHEP-SEIMC; Grupo de Estudio de Hepatitis Virica, of the Sociedad Andaluza de Enfermedades Infecciosas y Microbiologia Clinica: HEPAVIR / Red de Investigacion en SIDA (RIS-HEP07). Week 4 response predicts sustained virological response to all-oral direct-acting antiviral-based therapy in cirrhotic patients with hepatitis C virus genotype 3 infection. Clin Microbiol Infect. 2017 Jun;23(6):409.e5-409.e8. doi: 10.1016/j.cmi.2016.12.034. Epub 2017 Jan 28. PMID 28137633
- [Result] Neukam K, Morano-Amado LE, Rivero-Juarez A, Mancebo M, Granados R, Tellez F, Collado A, Rios MJ, de Los Santos-Gil I, Reus-Banuls S, Vera-Mendez F, Geijo-Martinez P, Montero-Alonso M, Suarez-Santamaria M, Pineda JA. HIV-coinfected patients respond worse to direct-acting antiviral-based therapy against chronic hepatitis C in real life than HCV-monoinfected individuals: a prospective cohort study. HIV Clin Trials. 2017 May;18(3):126-134. doi: 10.1080/15284336.2017.1330801. PMID 28599618
- [Result] Alvarez-Ossorio MJ, Sarmento E Castro R, Granados R, Macias J, Morano-Amado LE, Rios MJ, Merino D, Alvarez EN, Collado A, Perez-Perez M, Tellez F, Martin JM, Mendez J, Pineda JA, Neukam K; HEPAVIR-DAA, GEHEP-MONO, RIS-HEP07 and RIS-HEP13 Study Groups. Impact of interferon-free regimens on the glomerular filtration rate during treatment of chronic hepatitis C in a real-life cohort. J Viral Hepat. 2018 Jun;25(6):699-706. doi: 10.1111/jvh.12867. Epub 2018 Feb 27. PMID 29377515
- [Derived] Gonzalez-Serna A, Corma-Gomez A, Tellez F, Corona-Mata D, Rios-Villegas MJ, Merino D, Galera C, Collado-Romacho AR, De Los Santos I, Cucurull J, Santos M, Garcia-Martin S, Rivero A, Real LM, Macias J. Response to glecaprevir/pibrentasvir in HIV/HCV-coinfected patients in clinical practice. J Antimicrob Chemother. 2023 Oct 3;78(10):2591-2596. doi: 10.1093/jac/dkad278. PMID 37671831
- [Derived] Macias J, Morano LE, Tellez F, Granados R, Rivero-Juarez A, Palacios R, Rios M, Merino D, Perez-Perez M, Collado A, Figueruela B, Morano A, Freyre-Carrillo C, Martin JM, Rivero A, Garcia F, Pineda JA; HEPAVIR group from the Sociedad Andaluza de Enfermedades Infecciosas (SAEI) and the GEHEP group from the Sociedad Espanola de Enfermedades Infecciosas y Microbiologia (SEIMC). Response to direct-acting antiviral therapy among ongoing drug users and people receiving opioid substitution therapy. J Hepatol. 2019 Jul;71(1):45-51. doi: 10.1016/j.jhep.2019.02.018. Epub 2019 Mar 8. PMID 30853642